CLINICAL TRIAL: NCT01209845
Title: Low Dose Ketamine for Low Mood States: An Emergency Department Feasibility Study for Depressed Patients
Brief Title: Ketamine for Low Mood States in the ER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0909005766
Record Dates: First submitted 2010-08-30; First posted 2010-09-27 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Depression; Suicide Ideation
Keywords: depression; suicide ideation; emergency department; ketamine
MeSH Terms: conditions — Depression; Emergencies | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketamine (Experimental): Patients were administered a single sub-anaesthetic i.v. bolus of ketamine (0.2 mg/kg over 1-2 min) in the ED, with continuous monitoring of vital signs, adverse events and psychotomimetic side-effects for 4 h post-administration.
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine — intravenous ketamine(0.2 mg/kg) over 1-2 minutes IV

SUMMARY:
The investigators hope to see if a commonly used drug such as ketamine could help depressed ER patients feel better and improve their mood quickly.

DETAILED DESCRIPTION:
Rapid-onset antidepressants could have important clinical impact if their benefits extended to Emergency Department (ED) patients. We hope to explore the preliminary feasibility, tolerability and efficacy of single-dose, intravenous (IV) ketamine in depressed ED patients who presented with suicide ideation (SI).

The manuscript (article) for this study has been retracted because Yale University conducted an investigation that determined that the description of the research was not accurate. The article misrepresents both the protocol-specified doses and the actual delivered doses of ketamine.

ELIGIBILITY:
Inclusion Criteria:

* adults (>18yrs) presenting to the Emergency department with symptoms of depression and/or suicide ideation (MADRS>30) with ability to give informed consent.
* medically stable

Exclusion Criteria:

* psychosis, bipolar, or other significant physical or mental illness
* pregnancy
* non-voluntary status
* urine drug screen positive for drugs of abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | 40, 80, 120, 240 minutes after administration of drug
  The MADRS measures mood (depression) and item 10 measures suicide ideation.

SECONDARY OUTCOMES:
recruitment success and retention of subjects in the ER | initial recruitment of eligible subjects in the ER and for two weeks after administration of drug
  All patient subjects are admitted and we will follow them in the hospital and for 2 weeks after hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory L Larkin, MD, Principal Investigator — Yale University School of Medicine, Department of Emergency Medicine
Locations (1):
- Yale New Haven Hospital Emergency Department, New Haven, Connecticut, United States

REFERENCES:
- [Result] Larkin GL, Beautrais AL. A Preliminary Naturalistic Study of Low-Dose Ketamine for Depression and Suicide Ideation in the Emergency Department. Int J Neuropsychopharmacol. 2017 Jul 1;20(7):611. doi: 10.1093/ijnp/pyx035. No abstract available. PMID 28637184
- [Result] Larkin GL, Beautrais AL. A preliminary naturalistic study of low-dose ketamine for depression and suicide ideation in the emergency department. Int J Neuropsychopharmacol. 2011 Sep;14(8):1127-31. doi: 10.1017/S1461145711000629. Epub 2011 May 5. PMID 21557878 (Retraction: PMID 28637184 Int J Neuropsychopharmacol. 2017 Jul 1;20(7):611)